CLINICAL TRIAL: NCT05611255
Title: Comparison of Two Bladder Catheterization Strategies in Thoracic Surgery Patients With an Enhanced Recovery After Surgery (ERAS): Systematic Intermittent Catheterization Versus Bladder Scan Guided Catheterization in the Post Anesthesia Care Unit: a Prospective Randomized Double-blind Study
Brief Title: Comparison of Two Bladder Catheterization Strategies in Thoracic Surgery Patients With an Enhanced Recovery After Surgery (ERAS)
Acronym: URICATHOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety issue : increased occurrence of severe post-micturition residue (emergency urological consultation) for group B. The decision was taken on the advice of a committee of external experts
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RECHMPL20_0461
Record Dates: First submitted 2022-10-10; First posted 2022-11-10 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-05

CONDITIONS: Urinary Retention; Chronic Kidney Infection; Urinary Infection
Keywords: Urinary catheter; Acute urinary retention; Thoracic surgery; Thoracic epidural; Enhanced Recovery After Surgery (ERAS); Perioperative medicine
MeSH Terms: conditions — Urinary Retention; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic Intermittent Catheterization (SIC) (Experimental): A bladder catheter will be placed in the operating room, at the end of the operation, in a patient still under general anesthesia. Once the urine has been drained and quantified, the bladder catheter will be removed before the patient is discharged and extubated.
  Interventions: Procedure: Systematic Intermittent Catheterization
- Bladder Scan Guided Catheterization (BSGC) (Active Comparator): No systematic catheterization will be performed, the indication for catheterization will be guided by bladder-scan volume monitoring.
  Interventions: Procedure: Bladder Scan Guided Catheterization

INTERVENTIONS:
Procedure: Systematic Intermittent Catheterization — A strategy that consists of draining urine only once, in all patients, after surgery (in the operating room).
  Other Names: SIC
  Arms: Systematic Intermittent Catheterization (SIC)
Procedure: Bladder Scan Guided Catheterization — A strategy of standardized and reproducible assessment of bladder volume before discharge from the post anesthesia care unit, and draining urine only in patients who require it.
  Other Names: BSGC
  Arms: Bladder Scan Guided Catheterization (BSGC)

SUMMARY:
General anesthesia, thoracic epidural, and morphine inhibit the urination process and promote postoperative Acute Urinary Retention (AUR) after thoracic surgery. Indwelling bladder catheterization prevents this risk, but is associated with other complications (urinary tract infection, delayed mobilization). With the rise of enhanced recovery after surgery (ERAS) protocols, bladder catheterization is being questioned. The current protocol in the department is to catheterize only patients with a high bladder volume in the post anesthesia care unit (defined as a bladder volume > 400 ml on bladder scan). Preliminary results from the "AirLeaks" study show a high rate of early postoperative AUR (approximately 50%). The investigators believe that a "systematic intermittent catheterization" (SIC) strategy is superior to the current "bladder scan-guided catheterization in the post anesthesia care unit" (BSGC) strategy in preventing the risk of postoperative AUR. To their knowledge, no study has compared these two bladder catheterization strategies in a thoracic accelerated rehabilitation protocol.

DETAILED DESCRIPTION:
Acute urinary retention (AUR) is clinically defined by the presence of a bladder globe, with complete inability to urinate, sometimes associated with severe suprapubic abdominal pain. It is a urological emergency. An AUR can be complicated by acute renal failure, obstruction lifting syndrome (polyuria), a vacuo hematuria, or a slammed bladder (characterized by the presence of a post-void residue).

Systematic intermittent catheterization (SIC) allows monitoring of diuresis during the per- and post-operative period, and prevents the risk of AUR. It is associated with numerous disadvantages, such as the risk of infection (nosocomial urinary tract infection, bacteriuria, candiduria), which doubles after 2 days of catheterization, the risk of trauma (bleeding from the urethra, hematuria), the delay in mobilization and ambulation, and the psychological impact on the patients (dependence, agitation, confusion). All of these complications are potentially at risk of lengthening the average length of stay, and represent an additional cost for the Health Insurance. Thus, it seems that SIC is an obstacle to enhance recovery after surgery (ERAS), which is why the investigators have eliminated this option in our center. However, even recent American protocols for thoracic ERAS consider that an epidural should be associated with an indwelling catheter.

Bladder catheterization strategies are available for patients undergoing lung surgery. Options include no bladder catheterization, evacuation catheterization, and post anesthesia care unit catheterization guided by ultrasound or bladder scan measurement of bladder volume.

SIC is a strategy that involves draining urine once, in all patients, after surgery (in the operating room). Bladder Scan Guided Catheterization in the post anesthesia care unit (BSGC) is an innovative strategy that consists of a standardized and reproducible assessment of the bladder volume before discharge from the post anesthesia care unit, and draining urine only in patients who require it.

To their knowledge, no study has compared these two bladder catheterization strategies in a thoracic ERAS protocol.

The hypothesis is that a SIC strategy is superior to an individualized BSGC strategy in preventing postoperative AUR in thoracic surgery patients entering a ERAS program.

The SIC strategy is a novel idea that is not yet widely used in ERAS programs. The investigators believe that the SIC strategy will significantly decrease the rate of AUR. If this strategy proves to be superior to our current "bladder scan guided" service protocol, it could be incorporated into our ERAS program. Knowing the clinical repercussions, psychological impact, and costs associated with postoperative AUR, the medico-economic prospects of this study are major.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing scheduled thoracic surgery at the study center
* Be of legal age
* Be eligible for the enhanced recovery after surgery (ERAS) protocol in effect in the department.

Exclusion Criteria:

* Non-intubated anesthesia with spontaneous ventilation (NIVATS)
* Already have an indwelling bladder catheter or suprapubic catheter or double J catheter or other urinary drainage device
* Urinary tract infection under treatment or bladder catheterization less than one month old
* Indication of per- or postoperative bladder catheterization for another reason (e.g. monitoring of diuresis in chronic renal failure)
* Known vesico-sphincter disorder with documented post-void residue
* Neurological bladder (spinal cord injury or stroke sequelae)
* Documented urinary incontinence
* Chronic renal failure with a glomerular filtration rate (GFR) < 30 ml/min
* Contraindication to bladder catheterization (e.g. stenosis of the urethra)
* Be under legal protection or incapable of giving consent
* Failure to obtain written informed consent after a reflection period
* Not be affiliated to a French social security system or a beneficiary of such a system
* Long-term morphine drugs
* Pregnancy in progress or planned during the study period, Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of acute urinary retention (AUR) within 24 hours postoperatively | 24 hours after thoracic surgery
  AUR is defined by the absence of voiding recovery in an unprobed patient, with or without pubic pain (pain may be inhibited by epidural or morphine received), associated with a bladder volume > 400 ml on bladder scan.

SECONDARY OUTCOMES:
Occurrence of acute urinary retention (AUR) after Day 1 and during the first 5 days after surgery or during the hospital stay | Between Day 1 and Day 5 postoperative
  Compare the rate of AUR occurring beyond the 24th postoperative hour between the two groups.
Bladder volume drained | The first hour after catheter placement
  Bladder volume drained the first hour after catheter placement
Total duration of the first bladder catheterization | During the first bladder catheterization
  Total duration of the first bladder catheterization
Total number of bladder catheterizations | During the 5 days of post-surgical hospitalization
  Total number of bladder catheterizations
The rate of complications related to catheterization | During the 5 days of post-surgical hospitalization
  Macroscopic hematuria, documented urinary tract infection, suspected urinary tract infection with probabilistic antibiotic treatment.
The rate of complications related to AUR | During the 5 days of post-surgical hospitalization
  Postoperative acute renal failure
Other postoperative complications | During the 5 days of post-surgical hospitalization
  Postoperative hypotension, nausea or vomiting.
Duration before putting in the chair (in hours) | During the 5 days of post-surgical hospitalization
  Duration before putting in the chair (in hours)
Duration before standing up (in hours) | During the 5 days of post-surgical hospitalization
  Duration before standing up (in hours)
Length of hospital stay | During the 5 days of post-surgical hospitalization
  Length of hospital stay
Estimated cost of stay | During the 5 days of post-surgical hospitalization
  Estimated cost of stay

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No